CLINICAL TRIAL: NCT04570319
Title: A Randomized, Double Blind and Placebo-Controlled Clinical Trial to Evaluate the Effect of a Probiotic in Patients With Acne
Brief Title: Clinical Trial to Evaluate the Effect of a Probiotic in Acne
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bionou Research, S.L. (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ACNE.PROBI
Record Dates: First submitted 2020-04-16; First posted 2020-09-30 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Acne; Acne Vulgaris
Keywords: Probiotic; Acne; Microbiome; Microbiota; Symbiotic
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic Bths-08 (Experimental): a capsule containing the probiotic blend (nutritional complement)
  Interventions: Dietary Supplement: Probiotic Bths-08
- Placebo (Placebo Comparator): a capsule containing placebo comparator
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic Bths-08 — A capsule containing the probiotic blend (dietary supplement), administered once daily for 12 weeks
  Arms: Probiotic Bths-08
Dietary Supplement: Placebo — A capsule containing the placebo (dietary supplement), administered one daily for 12 weeks
  Arms: Placebo

SUMMARY:
A 12-week randomized, multicenter and double-blind, placebo-controlled study to evaluate the effect of a probiotic in the clinical and subjective evolution of acne in adolescent and adult patients.

DETAILED DESCRIPTION:
Acne is a chronic inflammatory disease of the skin that affects 85% of younger adults in westernized populations. Acne pathophysiology is multifactorial and may include alterations of the pilosebaceous unit function, skin microbiota, hormone imbalance and gut microbiota. Acne pathology shares features with inflammatory chronic conditions such as metabolic syndrome, obesity or diabetes.

Probiotics are live microorganisms that when administered in adequate amounts confer a health benefit for the host. Probiotics are proposed for the treatment of inflammatory chronic conditions, including dermatological diseases as atopic dermatitis and psoriasis. However, the clinical evidence is limited. Therefore, usefulness of probiotics for acne vulgaris treatment must be ascertained in humans.

This randomized study aims to evaluate the effect of a probiotic on the treatment and clinical and subjective evolution of acne vulgaris.

ELIGIBILITY:
Inclusion Criteria:

* Signature of informed consent by the patient (and their legal guardian in case of being under age).
* Age between 12 and 30 years-old.
* AGSS (Acne Global Severity Scale) Score: 2 or higher
* Patients who agree to follow the study's dietary recommendations.

Exclusion Criteria:

* Contraindication of any of the components of the product under study.
* Topical or systemic use of antifungals and antibiotics in the previous 2 weeks.
* Consumption of probiotics in the previous 2 months.
* Use of systemic retinoids in the previous 6 months.

Ages: 12 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 81 (Actual)
Dates: Start 2020-04-29 (Actual); Primary Completion 2022-07-21 (Actual); Study Completion 2022-09-20 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the AGSS (Acne Global Severity Scale) index at 12 weeks | 0 and 12-week
  Score between 0 and 5:
  0: Clean = Normal and clear skin without evidence of acne
  1. Almost clean = There are some non-inflammatory lesions, with uncommon and non-inflamed papules
  2. Mild = few inflammatory lesions (no nodule-cystic lesions)
  3. Moderate = Noninflammatory lesions predominate, but multiple inflammatory lesions appear (nodule-cystic lesions may be present)
  4. Severe = Inflammatory lesions predominate (nodule-cystic lesions may be present)
  5. Very severe = Highly inflammatory lesions predominate (several nodule-cystic lesions)
  Patients who improve in at least one category of the scale are considered as responders to treatment.

SECONDARY OUTCOMES:
Change from baseline in the number of acne lesions at week 12 | 0 and 12-week
  Number of non-inflammatory, inflammatory and total acne lesions.
Change from baseline in the GAGS (Global Acne Grading System) index at week 12 | 0 and 12-week
  TOTAL SCORE = [Nose S x 1 + Chin S x 1 + Front S x 2 + Right cheek S x 2 + Left cheek S x 2 + Torso S x 3]
  [Severity (S): 0 = Absence; 1 = Comedones; 2 = Papules; 3 = Pustules; 4 = Nodules]
  SCORE: 0 = Clean; 1-19 = Mild; 20-30 = Moderate; 31-38 = Severe; > 38 = Very severe
  Patients who have a reduction in the score of at least 30% are considered as responders to treatment.
Use of antibiotic acne treatment | 12-week
  Days of antibiotic use for the acne treatment, registered by the patient.
Change from the baseline in the patient subjective evaluation index at week 12 | 0 and 12-week
  Min score (Best) = 6 Max score (Worst) = 30
Change in the percentage of patients with presence of Cutibacterium acnes and Staphylococcus aureus in skin microbiome | 0 and 12-week
  Skin sample and genomic and microbiological analysis.
Adherence to treatment | 12-week
  Compliance rate (in percentage) calculated as the number of leftover capsules divided by the total number of days between visits.
Treatment safety assessed by number of adverse events | 12-week
  Number of adverse events that occur during the treatment period.

CONTACTS AND LOCATIONS:
Overall Officials: Vicente Navarro-Lopez, PhD; MD, Principal Investigator — Universidad Católica San Antonio de Murcia (UCAM)
Locations (4):
- Spain (4):
  - Universidad Católica San Antonio de Murcia, Guadalupe, Murcia
  - Centro Dermatológico Estético de Alicante, Alicante
  - Hospital Universitari Sagrat Cor, Barcelona
  - Clínica Eguren Dermatología y Estética, Madrid